CLINICAL TRIAL: NCT07138040
Title: Re-Engaging AYA Survivors in Cancer-Related Healthcare: A Sequential Multiple Assignment Randomized Trial
Brief Title: Re-Engaging AYA Survivors in Cancer-Related Healthcare
Acronym: REACH:SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Nationwide Children's Hospital (Other); University of Pennsylvania (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 22-020668; R01CA273328 (NIH)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Survivor; Adolescents and Young Adults; Digital Health Intervention; Adaptive Intervention; Sequential Multiple Assignment Randomized Trial; Long Term Follow Up Care; Survivorship Care Plan
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial with 2 stages of randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Written Intervention + Written Intervention (Responders) (Experimental): Start with written intervention (WI) in stage 1, those who respond (schedule an appointment) in stage 1 continue receiving WI in stage 2 (maintenance).
  Interventions: Behavioral: Stage 1 Written Information; Behavioral: Stage 2 Written Information
- Written Intervention + Low Touch Intervention (Responders) (Experimental): Start with written intervention (WI) in stage 1, those who respond (schedule an appointment) in stage 1, step up to receive low touch intervention (LTI) in stage 2.
  Interventions: Behavioral: Stage 1 Written Information; Behavioral: Stage 2 Low Touch Intervention
- Written Intervention + Low Touch Intervention (Non-Responders) (Experimental): Start with written intervention (WI) in stage 1, those who don't respond (do no schedule an appointment in stage 1), step up to receive low touch intervention (LTI) in stage 2.
  Interventions: Behavioral: Stage 1 Written Information; Behavioral: Stage 2 Low Touch Intervention
- Written Intervention + High Touch Intervention (Non-Responders) (Experimental): Start with written intervention (WI) in stage 1, those who don't respond (schedule and appointment) in stage 1, step up (maximum) to receive high touch intervention (HTI) in stage 2.
  Interventions: Behavioral: Stage 1 Written Information; Behavioral: Stage 2 High Touch Intervention
- Low Touch Intervention + Low Touch Intervention (Responders) (Experimental): Start with low touch intervention (LTI) in stage 1, those who respond (schedule an appointment in stage 1), continue receiving LTI in stage 2 (maintenance).
  Interventions: Behavioral: Stage 1 Low Touch Intervention; Behavioral: Stage 2 Low Touch Intervention
- Low Touch Intervention + High Touch Intervention (Responders) (Experimental): Start with low touch intervention (LTI) in stage 1, those who respond (schedule an appointment in stage 1), step up to receive high touch intervention (HTI) in stage 2.
  Interventions: Behavioral: Stage 1 Low Touch Intervention; Behavioral: Stage 2 High Touch Intervention
- Low Touch Intervention + High Touch Intervention (Non-Responders) (Experimental): Start with low touch intervention (LTI) in stage 1, those who don't respond (don't schedule an appointment) in stage 1, step up to receive high touch intervention (HTI) in stage 2.
  Interventions: Behavioral: Stage 1 Low Touch Intervention; Behavioral: Stage 2 High Touch Intervention

INTERVENTIONS:
Behavioral: Stage 1 Written Information — Stage 1 WI: consists of a letter from the survivorship care team with information about long-term follow-up care and relevant contacts to schedule an appointment.
  Other Names: S1 WI
  Arms: Written Intervention + High Touch Intervention (Non-Responders); Written Intervention + Low Touch Intervention (Non-Responders); Written Intervention + Low Touch Intervention (Responders); Written Intervention + Written Intervention (Responders)
Behavioral: Stage 1 Low Touch Intervention — Stage 1 LTI: consists of the WI stage 1 letter, a copy of their treatment summary with instructions for creating their own survivorship care plan, and one text message per week with information to schedule a follow-up care appointment.
  Other Names: S1 LTI
  Arms: Low Touch Intervention + High Touch Intervention (Non-Responders); Low Touch Intervention + High Touch Intervention (Responders); Low Touch Intervention + Low Touch Intervention (Responders)
Behavioral: Stage 2 Written Information — Stage 2 WI: consists of a letter from the survivorship care team with information about what to expect at a long-term follow-up care appointment.
  Other Names: S2 WI
  Arms: Written Intervention + Written Intervention (Responders)
Behavioral: Stage 2 Low Touch Intervention — Stage 2 LTI: consists of the WI stage 2 letter, a copy of their treatment summary with instructions for creating their own survivorship care plan, and two to three non-tailored (generic) text messages per week related to scheduling an appointment, overcoming barriers to follow-up care, and health self-management.
  Other Names: S2 LTI
  Arms: Low Touch Intervention + Low Touch Intervention (Responders); Written Intervention + Low Touch Intervention (Non-Responders); Written Intervention + Low Touch Intervention (Responders)
Behavioral: Stage 2 High Touch Intervention — Stage 2 HTI: consists of personalized mobile-friendly dashboard containing the WI letters, their treatment summary, survivorship care plan, and a growing discover section with helpful tailored resources. They will also receive four to six text messages per week with personalized messages related to their chosen health goal, personal barriers to attending cancer-related follow-up care, treatment-related risks, information about scheduling their long-term follow-up appointments, health self-management, and fun texts consisting of celebrity quotes, memes, and altruistic messages.
  Other Names: S2 HTI; HTI
  Arms: Low Touch Intervention + High Touch Intervention (Non-Responders); Low Touch Intervention + High Touch Intervention (Responders); Written Intervention + High Touch Intervention (Non-Responders)

SUMMARY:
The goal of this clinical trial is to test the efficacy (how well they work) of different digital interventions that deliver information to adolescent and young adult (AYA) survivors of childhood cancer to promote re-engagement in cancer-related long-term follow-up care (LTFU). The main aims are:

* To test the efficacy of adaptive interventions (AIs) that begin with low touch intervention (LTI) as compared to written information (WI) on attending an appointment, and self-reported self-management among AYA.
* To identify the most efficacious second-stage strategy for those who initially schedule/attend an appointment (maintenance vs. step-up) and for those who do not (step-up vs. step-up maximum).
* To assess multilevel factors contributing to the effects of re-engaging AYA and how best to integrate AIs into practice.

Throughout the duration of the study, participants will complete four surveys, receive a series of interventions, and may be asked to participate in an interview (post-intervention).

DETAILED DESCRIPTION:
Over 80% of children diagnosed with cancer become long-term survivors; however, 70% develop chronic or life-threatening late effects from treatment, and these often emerge during young adulthood. Guidelines recommend annual long-term follow-up care (LTFU) to manage and monitor for late effects, recurrence, or new cancer(s). Yet, as risk for late effects increases in young adulthood and survivors transition into adult-focused care, engagement in care plummets. Disengagement from LTFU leaves adolescent and young adult survivors (AYA) vulnerable to delayed or poorly managed diagnoses and relates to lower knowledge and self-management abilities. Thus, interventions targeting re-engagement of AYA are critical for this vulnerable population. The REACH (Re-Engaging AYA survivors in Cancer-related Healthcare) study will test a low touch intervention (LTI), consisting of reminder "nudge" text messages and informational resources for up to 4 weeks compared to an enhanced usual care group that will receive written information (WI) only.

In Stage 2, AYA will be re-randomized based on responsiveness to Stage 1 (i.e., whether or not they made an appointment) into 16 weeks of intervention. Responders will either be re-randomized to receive a continued intervention (maintenance) or a stepped-up condition, while non-responders will only receive a stepped-up condition. Step-up may include expanded LTI (more text messages) or a high touch intervention (HTI). The HTI includes text messages and digital resources, including a personalized survivorship care plan (SCP), and a mobile-friendly platform with information tailored to variables such as barriers to care, treatment history and recommendations, and a personal health goal. Additionally, social worker and/or nurse support will be available to help overcome barriers (e.g., access care).

The intervention options in Stage 2 are intended to enhance self-management beyond simply attending LTFU in order to sustain long-term engagement. Outcomes are measured after Stage 1 (T2), Stage 2 (T3) and at 36 weeks (T4).

It is expected that those who start with LTI versus WI will be more likely to attend a LTFU appointment by T4. For Stage 2, those who receive the stepped-up condition compared to those with maintenance, and those who received HTI compared to LTI, will be more likely to attend an appointment by T4. Attending an appointment by T3 and indices of self-management are secondary outcomes. The study team will assess moderators of intervention outcomes, intervention engagement, acceptability, feasibility, and cost. Qualitative interviews will assess multilevel barriers and facilitators of future implementation with stakeholders (AYA, parents/supports, providers, administrators). This trial aims to promote optimal engagement in LTFU and self-management for AYA survivors, improving outcomes and reducing disparities. For Stage 2, those who receive the stepped-up condition compared to those with maintenance, and those who received HTI compared to LTI, will be more likely to attend an appointment by T4.

ELIGIBILITY:
Inclusion Criteria for AYA

1. 15-29 years old
2. History of a childhood cancer diagnosis, diagnosed prior to age 22
3. Has not had a cancer-related follow-up visit in at least 15 months (or is 3 months past recommended follow-up)
4. U.S. resident (not international patient)
5. Has previously attended a cancer-related appointment at Children's Hospital of Philadelphia, or Nationwide Children's Hospital or Penn
6. At least 2 years from end of treatment and 5 years from diagnosis
7. English proficient
8. For AYA under age 18, must have a caregiver to provide informed consent

Exclusion Criteria for AYA

1. Cognitive impairment limiting participation
2. Received surgery only treatment
3. Transferred to primary care
4. Currently living with cancer diagnosis (either new, metastatic, recurrence, or relapse)
5. Absence of documentation of treatment history
6. Absence of inclusion criteria above

Inclusion Criteria for Support Person of AYA

1. Primary caregiver or other support person (e.g. partner, sibling, other caregiver)
2. At least 18 years old
3. U.S. resident
4. English proficient

Exclusion Criteria for Support Person of AYA

1. No involvement in the AYA's healthcare
2. AYA Decline support person's participation
3. Absence of inclusion criteria above

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Re-Engagement in Care - by T4 | 36 weeks (T4)
  Percentage of participants who re-engage in care (attend a LTFU appointment) by T4 as measured by electronic health record (EHR) review. If attendance is not viewable in EHR, it will be ascertained by self-report (yes/no).

SECONDARY OUTCOMES:
Re-Engagement in Care - by T3 | 20 weeks (T3)
  Percentage of participants who re-engage in care (attend a LTFU appointment) by T3 as measured by electronic health record (EHR) review. If attendance is not viewable in EHR, it will be ascertained by self-report (yes/no).
AYA Self-Management (Health Knowledge Inventory) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Health Knowledge inventory (28 items), a total percentage correct score will be reported 0-100%, with higher scores representing greater self-management.
AYA Self-Management (Transition Readiness Questionnaire) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Transition Readiness Assessment Questionnaire (20 items), a total average score will be reported ranging from 1-5, with higher scores representing greater self-management.
AYA Self-Management (Self-Management Skills) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Self-management Skills Scale (15 items), a total percentage score will be reported ranging from 0-100%, with higher scores representing greater self-management.
AYA Self-Management (Health Goal Progress) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Health Goal Progress (5 items), a total score will be reported ranging from 5-24, with higher scores representing greater self-management.
AYA Self-Management (Allocation of Treatment Responsibility) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Allocation of treatment responsibility, clinic appointment subscale (5 items), a total score will be reported ranging from 5-20, with higher scores representing greater self-management.
AYA Self-Management (Transition Readiness Inventory) | 2 times - at 20 weeks (T3) and 36 weeks (T4)
  Measured via self-reported participant questionnaire. For the Transition Readiness Inventory (28 items), a total average score will be reported ranging from 1-5, with higher scores representing greater self-management.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Penn Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided